CLINICAL TRIAL: NCT00991809
Title: A Pilot Study of Prolonged, Intermittent Exposure to Alfentanil on Opioid-Induced Hyperalgesia in Healthy Volunteers
Brief Title: Study on the Development of Opioid Induced Hyperalgesia (OIH) After Exposure to Alfentanil
Acronym: 0813
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NA_00022154; 1K24DA023186 (NIH)
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-09

CONDITIONS: Hyperalgesia
Keywords: opioid induced hyperalgesia
MeSH Terms: conditions — Hyperalgesia | interventions — Alfentanil; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alfentanil (Experimental): Subjects received a series of acute alfentanil administrations each session (15 mcg/kg IM per session), with sessions spaced at 3-4 day intervals.
  Interventions: Drug: Alfentanil
- Diphenhydramine (Active Comparator): Subjects received a series of acute diphenhydramine administrations each session (25 mg IM per session), with sessions spaced at 3-4 day intervals.
  Interventions: Drug: Diphenhydramine

INTERVENTIONS:
Drug: Alfentanil — 15 mcg/kg IM
  Arms: Alfentanil
Drug: Diphenhydramine — 25 mg IM
  Other Names: Benadryl
  Arms: Diphenhydramine

SUMMARY:
The purpose of this study was to follow a person's response to experimental pain after multiple consecutive exposures to alfentanil or diphenhydramine to see if the person can tolerate the pain more, less, or the same at the end of the study.

DETAILED DESCRIPTION:
This project investigates the phenomenon of opioid-induced hyperalgesia (OIH). Opioid analgesics, in addition to their therapeutic anti-nociceptive effects, under some conditions produce pro-nociceptive effects. This phenomenon of pain or pain sensitivity being increased by prior opioid administration is called opioid-induced hyperalgesia. It is thought to be relevant both to pain management complications and to complications of opioid dependence and its treatment. This study investigated the time-course of opioid-induced hyperalgesia development in healthy normal volunteers (N=12 completers), using a series of acute alfentanil administrations (15 mg/kg mg intramuscular (IM) per day) spaced at 3-4 day intervals, with testing for pain tolerance using the cold pressor test (CPT), and mechanical quantitative sensory testing (MQST) each administered repeatedly over time within each testing day. The goal was to determine the time course of OIH development following acute opioid administration, and to assess whether this changes over repeated acute opioid administrations.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55
* No active medical conditions
* BMI between 20-30
* Able and willing to perform/tolerate pain procedures
* Able to communicate in English

Exclusion Criteria:

* Lifetime substance use disorder, except for alcohol abuse/dependence in remission
* Use of opiates in last 3 months
* Ongoing marijuana use
* Acute or chronic pain
* Neurologic or psychiatric condition known to influence cold pressor testing (peripheral neuropathy, major depression, or schizophrenia)
* Current use of prescribed or over the counter pain medications
* Previous adverse reaction to opiate medications or diphenhydramine
* Use of tobacco or caffeine on study days

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Tompkins, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Result] Tompkins DA, Smith MT, Bigelow GE, Moaddel R, Venkata SL, Strain EC. The effect of repeated intramuscular alfentanil injections on experimental pain and abuse liability indices in healthy males. Clin J Pain. 2014 Jan;30(1):36-45. doi: 10.1097/AJP.0b013e3182851758. PMID 23446076

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment began in February 2009 after Institutional Review Board (IRB) approval. Screening started on 2/9/09. The last person was screened on 3/12/2010 and finished the study in April 2010. A total of 42 screenings occurred and 12 persons completed the study. Recruitment was conducted at the Behavioral Pharmacology Research Unit (BPRU).
Pre-assignment Details: Since study initiation in February 2009, there were 42 persons consented. There were 13 screen failures [4 had urines positive for illicit substances, 4 had BMI>30, 5 had active medical problems]. Seven met study criteria but decided not to start as they could not commit to study schedule (N=6) or did not like blood draws (N=1)
Groups:
- Alfentanil: Subjects received a series of acute alfentanil administrations each session (15 mcg/kg IM per session), with sessions spaced at 3-4 day intervals.
  Alfentanil : 15 mcg/kg intramuscular(IM)
- Diphenhydramine: Subjects received a series of acute diphenhydramine administrations each session (25 mg IM per session), with sessions spaced at 3-4 day intervals.
  Diphenhydramine : 25 mg IM
Period: Overall Study
Arm/Group | Alfentanil | Diphenhydramine
Started | 12 | 10
Completed | 8 | 4
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Alfentanil: These subjects will receive a series of acute alfentanil administrations each session (15 mcg/kg IM per session), with sessions spaced at 3-4 day intervals.
  Alfentanil : 15 mcg/kg IM
- Diphenhydramine: Subjects will receive a series of acute diphenhydramine administrations each session (25 mg IM per session), with sessions spaced at 3-4 day intervals.
  Diphenhydramine : 25 mg IM
- Total: Total of all reporting groups
Arm/Group | Alfentanil | Diphenhydramine | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 10 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Pain Tolerance
Description: The participant places their hand in a water bath kept at 4 degrees Celsius (cold pressor test). They then continue to hold the hand in the water bath until they can no longer tolerate the pain (pain tolerance) or until the end of the testing (truncated at 300 seconds for safety purposes). Reported as the mean (time to hand removal in seconds) at the 30 minute time point.
Time Frame: 8 sessions over 4-6 weeks
Population: One person in the diphenhydramine group was dropped from analysis, even though he completed the study as he tolerated cold pressor testing for the maximum amount of time in sessions 2-8.
Measure: Mean (Full Range); unit: seconds
Arm/Group | Alfentanil | Diphenhydramine
Number analyzed (Participants) | 8 | 3
seconds | 105.3 [10.5 to 300] | 19.2 [7.1 to 38.7]

2. Secondary Outcome: Pain Threshold
Description: The amount of time (in seconds) before the participant first verbally reports feeling pain after placing hand in 4 degree Celsius circulating water bath at the 30 minute time point. Truncated at 300 seconds for safety purposes.
Time Frame: 8 sessions over 4-6 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: seconds
Groups:
- Alfentanil: These subjects will receive a series of acute alfentanil administrations each session (15 mcg/kg IM per session), with sessions spaced at 3-4 day intervals.
  Alfentanil: 15 mcg/kg IM
- Diphenhydramine: Subjects will receive a series of acute diphenhydramine administrations each session (25 mg IM per session), with sessions spaced at 3-4 day intervals.
  Diphenhydramine: 25 mg IM
Arm/Group | Alfentanil | Diphenhydramine
Number analyzed (Participants) | 8 | 3
seconds | 20.7 [4.6 to 73.6] | 8.6 [4.4 to 22.5]

ADVERSE EVENTS:
Arm/Group | Alfentanil | Diphenhydramine
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/10

LIMITATIONS AND CAVEATS:
The sample size was intentionally small as this was to be a preliminary proof-of-concept step in the development of a human OIH model.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No